CLINICAL TRIAL: NCT00752726
Title: The Effects of Weight Reduction With Orlistat vs. Placebo on Changes in Body Composition
Brief Title: Effect of Orlistat in Body Composition
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: W3600586
Record Dates: First submitted 2008-09-11; First posted 2008-09-15 (Estimated); Results first posted 2013-02-07 (Estimated); Last update posted 2013-03-08 (Estimated); Status verified 2013-02

CONDITIONS: Obesity; Overweight
Keywords: overweight, orlistat, body composition
MeSH Terms: conditions — Obesity; Overweight | interventions — Orlistat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Orlistat (Active Comparator): Orlistat 60 milligram (mg) capsules to be consumed orally with each meal 3 times per day
  Interventions: Drug: Orlistat
- Placebo (Placebo Comparator): Placebo to match Orlistat 60 mg capsules to be consumed orally with each meal 3 times per day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Orlistat — Weight loss treatment
  Arms: Orlistat
Drug: Placebo — Inactive
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if a 24 week weight loss program with orlistat 60 mg will produce greater changes in body composition compared to placebo.

DETAILED DESCRIPTION:
Large amounts of VAT (adipose tissue surrounding the viscera of the organs), is known to be associated with increased risk of heart disease and diabetes. Orlistat (tetrahydrolipstatin or THL) inhibits gastrointestinal lipase and reduces the absorption of dietary fat. The purpose of this study is to to determine if a 24 week weight loss program with orlistat 60 mg would produce greater changes in adipose tissue depots (specifically VAT) compared to placebo. This study will use the Echo MRI technology across multiple sites to measure total fat mass. EchoMRI is a non invasive method ideally suited for studies which track changes in human body composition over time, with measuring times of less than 3 minutes and no radiation exposure.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-60 years inclusive
* Body Mass Index (BMI): BMI in the range of 25.0-34.9 kg/m^2
* Waist circumference:

Females: > 35 inches Males: > 40 inches

* Diet:

  1. Normal eating habits, consuming 3 meals a day (breakfast, lunch and dinner)
  2. Willing to follow a hypocaloric diet during the study to achieve weight loss
  3. Willing to take a daily multivitamin for the duration of the study.
* General Health:Good general health with (in the opinion of the investigator) no clinically significant and relevant abnormalities of medical history or physical examination

Exclusion Criteria:

* Pregnant and/ or Breast-feeding women
* Diet/Exercise:Currently on a special diet or who cannot fulfill the dietary requirements of the study.
* Smoking History:a) Smoking cessation within the past 6 months b) Current Smokers
* Allergy/Intolerance: Known or suspected intolerance or hypersensitivity to the study materials and study foods (or closely related compounds) or any of their stated ingredients.
* Medication:

  a) Currently taking medication for weight loss or appetite control. b) Previous Xenical® (orlistat) or alli® use within 3 months of screening date c) Currently taking medication or supplements that influence intestinal transit time and other stool formation parameters or influences cramping (e.g., Anticholinergics (such as atropine) or cholinergics (such as physostigmine), phenothiazines, tricyclic antidepressants, opioid analgesics (including loperamide), calcium channel antagonists, clonidine, cisapride, octreotide. Also, any laxative or antidiarrheal product). d) Currently taking or withdrawn during the past 6 months any drugs with significant impact on body weight (e.g. serotoninergically acting drugs, antidepressants, central adrenergically acting drugs, drugs inhibiting digestion and absorption, appetite suppressants, metformin) e) Currently taking Cyclosporine, Warfarin or Amiodarone HCL
* Disease/Surgery:

  a) History of gastrointestinal disease (e.g., irritable bowel syndrome, diarrhea, inflamed bowel, steatorrhea/fat malabsorption, hemorrhoids, incontinence, pancreatitis). b) History of psychological disorder, including eating disorders such as anorexia nervosa and bulimia c) History of neurological disorder (e.g. seizures, parkinson's disease, Alzheimer's disease) d) History of hypo/hyperthyroidism unless euthyroid and controlled on a stable dose of medication for at least 6 months. e) History of surgery for weight loss f) Uncontrolled hypertension g) Heart Disease h) Diabetes Mellitus (Type 1 and 2) (Fasting Blood Glucose >126 mg/dL)
* Participant has a known history of panic attacks and/or claustrophobia or other conditions precluding safe EchoMRI, CT or other scanning modalities according to local guidelines, (e.g., pacemaker, hearing aid, metallic body piercing and/or other metal implants) or in the opinion of the Investigator the participant exceeds size limitations for the instruments.
* Participant has had a weight loss or gain of greater than or equal to 3 kg in the 3 months prior to screening.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 131 (Actual)
Dates: Start 2008-09; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- United States (2):
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - Duke Clinical Research Unit, Durham, North Carolina
- Sahlgrenska Academy, Gothenburg, West Gothland, Sweden

REFERENCES:
- [Background] Smith SR, Stenlof KS, Greenway FL, McHutchison J, Schwartz SM, Dev VB, Berk ES, Kapikian R. Orlistat 60 mg reduces visceral adipose tissue: a 24-week randomized, placebo-controlled, multicenter trial. Obesity (Silver Spring). 2011 Sep;19(9):1796-803. doi: 10.1038/oby.2011.143. Epub 2011 Jun 30. PMID 21720429

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multicentric clinical study was conducted in 2 countries; 2 centres in United States of America (USA) and 1 centre in Sweden.
Pre-assignment Details: Out of 267 screened participants, 131 were randomized, while 136 participants were considered as screen failures.
Groups:
- Orlistat 60 Milligram (mg): Orlistat 60 mg capsules taken orally with meals 3 times per day
- Placebo: Placebo to match orlistat 60 mg capsules taken orally with meals 3 times per day
Period: Overall Study
Arm/Group | Orlistat 60 Milligram (mg) | Placebo
Started | 65 | 66
Safety Population | 63 (2 participants were never dosed with the study medication.) | 64 (2 participants were never dosed with the study medication.)
Intention to Treat (ITT) Population | 62 (ITT population had atleast 1 post treatment efficacy measurement.) | 61 (ITT population had atleast 1 post treatment efficacy measurement.)
Completed | 54 | 53
Not Completed | 11 | 13
Not completed — Lost to Follow-up | 2 | 1
Not completed — Adverse Event | 3 | 0
Not completed — Withdrawal by Subject | 5 | 10
Not completed — Other Reason | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Orlistat 60 mg: Orlistat 60 mg capsules taken orally with meals 3 times per day. Intent-to-treat (ITT) population was considered for baseline measures.
- Placebo: Placebo to match Orlistat 60 mg capsules taken orally with meals 3 times per day. ITT population was considered for baseline measures.
- Total: Total of all reporting groups
Arm/Group | Orlistat 60 mg | Placebo | Total
Number analyzed (Participants) | 62 | 61 | 123
Age Continuous [Mean (Standard Deviation); unit: Year] | 42.92 (9.031) | 43.84 (11.682) | 43.37 (10.397)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 51 | 102
  Male | 11 | 10 | 21
Body Weight [Mean (Standard Deviation); unit: Kilogram (kg)] | 88.10 (10.705) | 87.79 (9.354) | 87.95 (10.018)
Height [Mean (Standard Deviation); unit: Centimeter (cm)] | 168.30 (8.275) | 168.08 (8.117) | 168.19 (8.164)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kilogram per meter square (kg/m^2)] | 31.03 (2.259) | 31.04 (2.064) | 31.03 (2.155)
Waist Circumference [Mean (Standard Deviation); unit: cm] | 100.10 (7.967) | 100.60 (6.892) | 100.35 (7.427)
Visceral Abdominal Tissue (VAT) Mass [Mean (Standard Deviation); unit: kg] | 3.75 (1.870) | 3.92 (1.806) | 3.83 (1.832)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 24 in Abdominal VAT Mass
Description: VAT was measured by the computed tomography (CT) scan.
Time Frame: Baseline to week 24
Population: This analysis was carried out for the observed ITT population, who had this post-baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: kg
Groups:
- Orlistat 60 mg: Orlistat 60 mg capsules taken orally with meals 3 times per day
Arm/Group | Orlistat 60 mg | Placebo
Number analyzed (Participants) | 55 | 54
kg | -0.630 (0.6887) | -0.403 (0.7249)
Statistical Analysis 1: Comparison: Orlistat 60 mg vs Placebo; The null hypothesis considered no difference in the change from baseline to week 24 between the two treatment groups; Test type: Superiority or Other; p = 0.0244, ANCOVA — P-value was not adjusted for multiple comparisons; Mean change was adjusted for treatment, baseline VAT and center effect using an ANCOVA model; Adjusted Mean Difference = 0.263, 95% CI 2-sided [0.035 to 0.491], Standard Error of Mean 0.1150 — Adjusted mean difference between Placebo group and Orlistat group was determined. For this primary analysis, only one statistical test was performed and therefore, no multiple comparison adjustment was done

2. Secondary Outcome: Change From Baseline to Week 12 in Abdominal VAT Mass
Description: Abdominal VAT mass from baseline to week 12 was measured by CT scan.
Time Frame: Baseline to week 12
Population: This analysis was carried out for the observed ITT population, who had this post-baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Orlistat 60 mg | Placebo
Number analyzed (Participants) | 55 | 53
kg | -0.496 (0.4943) | -0.351 (0.5904)
Statistical Analysis 1: Comparison: Orlistat 60 mg vs Placebo; The null hypothesis considered no difference in the change from baseline to week 12 between the two treatment groups; Test type: Superiority or Other; p = 0.0415, ANCOVA — P-value was not adjusted for multiple comparisons; Mean change was adjusted for the treatment, baseline VAT and center effects using an ANCOVA model; Adjusted Mean Difference = 0.172, 95% CI 2-sided [0.007 to 0.337], Standard Error of Mean 0.0834 — Adjusted mean difference between Placebo group and Orlistat group was determined

3. Secondary Outcome: Change From Baseline to Week 24 in Body Weight
Description: Participants were weighed at least twice until two consecutive measurements were within 0.5 kg of each other and the average of the two measurements was recorded.
Time Frame: Baseline to week 24
Population: This analysis was carried out for the observed ITT population, who had this post-baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Orlistat 60 mg | Placebo
Number analyzed (Participants) | 54 | 53
kg | -5.96 (4.743) | -3.91 (5.375)
Statistical Analysis 1: Comparison: Orlistat 60 mg vs Placebo; The null hypothesis considered no difference in the change from baseline to week 24 between the two treatment groups; Test type: Superiority or Other; p = 0.026, ANCOVA — P-value was not adjusted for multiple comparisons; Mean change was adjusted for the treatment, baseline weight and center effects, using an ANCOVA model; Adjusted Mean Difference = 1.99, 95% CI 2-sided [0.25 to 3.74], Standard Error of Mean 0.881 — Adjusted mean difference between Placebo group and Orlistat group was determined

4. Secondary Outcome: Change From Baseline to Week 24 in Total Fat Mass
Description: Change in total fat mass was calculated from an average of three measurements at each visit from Echo Magnetic Resonance Imaging (EchoMRI).
Time Frame: Baseline to week 24
Population: This analysis was carried out for the observed ITT population, who had this post-baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Orlistat 60 mg | Placebo
Number analyzed (Participants) | 54 | 53
kg | -4.69 (3.691) | -3.16 (4.248)
Statistical Analysis 1: Comparison: Orlistat 60 mg vs Placebo; The null hypothesis considered no difference in the change from baseline to week 24 between the two treatment groups; Test type: Superiority or Other; p = 0.0242, ANCOVA — P-value was not adjusted for multiple comparisons; Mean change was adjusted for the treatment, baseline total fat mass and center effects using an ANCOVA model; Adjusted Mean Difference = 1.642, 95% CI 2-sided [0.219 to 3.065], Standard Error of Mean 0.7174 — Adjusted mean difference between placebo group and Orlistat group was determined

5. Secondary Outcome: Change From Baseline to Week 24 in Percentage Body Fat
Description: Body fat was assessed through Bioelectrical Impedance Analysis (BIA).
Time Frame: Baseline to week 24
Population: This analysis was carried out for the observed ITT population, who had this post-baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: Percentage (%) body fat
Arm/Group | Orlistat 60 mg | Placebo
Number analyzed (Participants) | 54 | 53
Percentage (%) body fat | -1.70 (3.434) | -0.38 (4.232)
Statistical Analysis 1: Comparison: Orlistat 60 mg vs Placebo; The null hypothesis considered no difference in the change from baseline to week 24 between the two treatment groups; Test type: Superiority or Other; p = 0.039, ANCOVA — P-value was not adjusted for multiple comparisons; Mean was adjusted for the treatment, baseline total fat mass and center effects using an ANCOVA model; Adjusted Mean Difference = 1.47, 95% CI 2-sided [0.07 to 2.87], Standard Error of Mean 0.704 — Adjusted mean difference between placebo group and Orlistat group was evaluated

6. Secondary Outcome: Change From Baseline to Week 24 in Waist Circumference
Description: Waist circumference was measured against the skin, without interference from clothing, at the level midway between the lateral lower rib margin and the iliac crest in standing position.
Time Frame: Baseline to week 24
Population: This analysis was carried out for the observed ITT population, who had this post-baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Orlistat 60 mg | Placebo
Number analyzed (Participants) | 54 | 53
cm | -6.65 (0.692) | -4.95 (0.704)
Statistical Analysis 1: Comparison: Orlistat 60 mg vs Placebo; The null hypothesis considered no difference in the change from baseline to week 24 between the two treatment groups; Test type: Superiority or Other; p = 0.085, ANCOVA — P-value was not adjusted for multiple comparisons; Mean change was adjusted for the treatment, baseline waist circumference and center effects, using an ANCOVA model; Adjusted Mean Difference = 1.70, 95% CI 2-sided [-0.24 to 3.63], Standard Error of Mean 0.974 — Adjusted mean difference between Placebo group and Orlistat group was determined

7. Secondary Outcome: Change From Baseline to Week 24 in Percentage Liver Fat
Description: For Liver fat, Intrahepatic lipids (IHL) were measured by Magnetic Resonance Spectroscopy (MRS).
Time Frame: Baseline to week 24
Population: ITT subset (participants who had this post-baseline efficacy assessment) from one study site was analysed for this parameter.
Measure: Mean (Standard Deviation); unit: Percentage (%) IHL
Arm/Group | Orlistat 60 mg | Placebo
Number analyzed (Participants) | 9 | 8
Percentage (%) IHL | -0.0008 (0.00609) | -0.0112 (0.03642)

8. Secondary Outcome: Change From Baseline to Week 24 in Liver Fat
Description: The liver fat was measured by CT scan in Hounsfield Units (HU).
Time Frame: Baseline to week 24
Population: This analysis was carried out for the observed ITT population, who had this post-baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: Hounsfield Units (HU)
Arm/Group | Orlistat 60 mg | Placebo
Number analyzed (Participants) | 54 | 53
Hounsfield Units (HU) | 0.06 (0.169) | 0.02 (0.174)
Statistical Analysis 1: Comparison: Orlistat 60 mg vs Placebo; The null hypothesis considered no difference in the change from baseline to week 24 between the two treatment groups; Test type: Superiority or Other; p = 0.3235, ANCOVA — P-value was not adjusted for multiple comparisons; Mean change was adjusted for the treatment, baseline liver fat and center effects, using an ANCOVA model; Adjusted Mean Difference = -0.023, 95% CI 2-sided [-0.069 to 0.023], Standard Error of Mean 0.0232 — Adjusted mean difference between placebo group and Orlistat group was evaluated

9. Secondary Outcome: Change From Baseline to Week 24 in Total Calories Expended for Physical Activity
Description: Measurement of physical activity from Paffenbarger questionnaire. The number of caloried expended was representation of activity level: Higher calorie counts indicate higher activity
Time Frame: Baseline to week 24
Population: This analysis was carried out for the observed ITT population, who had this post-baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: Kilocalorie (kcal)/week
Arm/Group | Orlistat 60 mg | Placebo
Number analyzed (Participants) | 54 | 53
Kilocalorie (kcal)/week | -498 (6627) | 517 (4873)
Statistical Analysis 1: Comparison: Orlistat 60 mg vs Placebo; The null hypothesis considered no difference in the change from baseline to week 24 between the two treatment groups; Test type: Superiority or Other; p = 0.28, ANCOVA — P-value was not adjusted for multiple comparisons; Mean change was adjusted for the treatment, baseline total calories expended and center effects using an ANCOVA model; Adjusted Mean Difference = 783.8, 95% CI 2-sided [-657.3 to 2224.9], Standard Error of Mean 726.54 — Adjusted mean difference between placebo group and Orlistat group was evaluated

10. Secondary Outcome: Change From Baseline to Week 24 in Quality of Life (QoL) Scores.
Description: QoL scores were measured using an Impact of Weight Quality of Life (IWQoL) Questionnaire, which scored the responses at a scale of 1 to 5(1, never true, to 5, always true): QoL scales for physical function, self-esteem, sexual life, public distress, and work were evaluated, and summarized in a total score. A higher value indicated a better quality of life.
Time Frame: Baseline to week 24
Population: This analysis was carried out for the observed ITT population, i.e. ITT subjects who had this post-baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Orlistat 60 mg | Placebo
Number analyzed (Participants) | 53 | 52
Score on a Scale | 5.29 (8.009) | 8.78 (10.429)
Statistical Analysis 1: Comparison: Orlistat 60 mg vs Placebo; The null hypothesis considered no difference in the change from baseline to week 24 between the treatment groups; Test type: Superiority or Other; p = 0.2847, ANCOVA — P-value was not adjusted for multiple comparisons; Mean difference was adjusted for the treatment, baseline value and center effects using an ANCOVA model; Adjusted Mean Difference = 1.66, 95% CI 2-sided [-1.40 to 4.72], Standard Error of Mean 1.542 — Adjusted mean difference was calculated as placebo minus orlistat

11. Secondary Outcome: Selectivity Index at Week 24
Description: The selectivity index (SI) was used as a measure of orlistat's ability to target abdominal VAT loss compared to total adipose tissue lost. SI was calculated using the following equation: Mean % change in VAT divided by Mean % change in total fat mass.
Time Frame: Baseline to week 24
Population: This analysis was carried out for the observed ITT population, who had this post-baseline efficacy assessment, only in Orlistat 60 mg group. This analysis was not carried out for placebo group.
Measure: Number; unit: Ratio
Arm/Group | Orlistat 60 mg
Number analyzed (Participants) | 54
Ratio | 1.155

ADVERSE EVENTS:
Time Frame: All adverse events encountered or spontaneously reported by the participant following administration of any investigational product (including washout product), or for up to 5 days after the last administration of investigational product
Arm/Group | Orlistat 60 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 2/63 | 1/64
Other Adverse Events (participants affected / at risk) | 57/63 | 52/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Orlistat 60 mg (N=63) | Placebo (N=64)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Biliary tract disorder (Hepatobiliary disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Orlistat 60 mg (N=63) | Placebo (N=64)
Fatty/oily stool (Gastrointestinal disorders) | 22 (36) | 3 (4)
Soft stools (Gastrointestinal disorders) | 14 (17) | 8 (10)
Flatulence (Gastrointestinal disorders) | 12 (16) | 5 (6)
Liquid stools (Gastrointestinal disorders) | 7 (8) | 5 (5)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 6 (8)
Increased defecation (Gastrointestinal disorders) | 6 (7) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 4 (5)
Fecal urgency (Gastrointestinal disorders) | 1 (2) | 4 (5)
Flatus with discharge (Gastrointestinal disorders) | 5 (5) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 1 (1)
Oily spotting (Gastrointestinal disorders) | 4 (4) | 0 (0)
Nasopharyngitis (Infections and infestations) | 25 (29) | 22 (33)
Gastroenteritis (Infections and infestations) | 2 (2) | 5 (7)
Influenza (Infections and infestations) | 5 (5) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3) | 4 (4)
Headache (Nervous system disorders) | 4 (5) | 4 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.